CLINICAL TRIAL: NCT03874026
Title: Cetuximab, Irinotecan and Fluorouracile in FiRst-line Treatment of Immunologically-selected Advanced Colorectal Cancer Patients: the CIFRA Study
Brief Title: Study of Folfiri/Cetuximab in FcGammaRIIIa V/V Stage IV Colorectal Cancer Patients
Acronym: CIFRA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 60/18
Record Dates: First submitted 2019-02-26; First posted 2019-03-14 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer; ADCC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Folfiri/Cetuximab (Experimental): Cetuximab 400 mg/mq intravenously (iv) with "load" dose of 400 mg/mq at the first cycle followed by 250 mg/mq iv weekly by iv infusion in 90 minutes. The administration of irinotecan will precede that of cetuximab and will consist on a dose of 180 mg/mq iv in 60 minutes every two weeks and it will be followed by fluorouracil (5-FU) at a dose of 400 mg/mq in slow iv bolus at half of lederfolin 200 mg/mq 2-hours infusion. At the end of the infusion of lederfolin an elastomeric pump loaded with 5-FU 2400 mg/mq in continuous 46 hours iv infusion will be applied. Only at the first administration of CT ("load" dose of cetuximab), irinotecan will not be administered.
  Interventions: Drug: Folfiri/Cetuximab

INTERVENTIONS:
Drug: Folfiri/Cetuximab — Cetuximab 400 mg/mq intravenously (iv) with "load" dose of 400 mg/mq at the first cycle followed by 250 mg/mq iv weekly by iv infusion in 90 minutes. The administration of irinotecan will precede that of cetuximab and will consist on a dose of 180 mg/mq iv in 60 minutes every two weeks and it will be followed by fluorouracil (5-FU) at a dose of 400 mg/mq in slow iv bolus at half of lederfolin 200 mg/mq 2-hours infusion. At the end of the infusion of lederfolin an elastomeric pump loaded with 5-FU 2400 mg/mq in continuous 46 hours iv infusion will be applied. Only at the first administration of CT ("load" dose of cetuximab), irinotecan will not be administered.

SUMMARY:
Patients' selection thorough the identification of predictive factors still represent a challenge in metastatic colorectal cancer (mCRC). Cetuximab (Erbitux®), a chimeric monoclonal antibody binding to the Epidermal Growth Factor Receptor (EGFR), belongs to the Immunoglobulins (Ig) grade 1 subclass able to elicit both in vitro and in vivo the Antibody-Dependent Cell-mediated Cytotoxicity (ADCC). ADCC is the cytotoxic killing of antibody-coated target cells by immunologic effectors. The effector cells express a receptor for the Fc portion of these antibodies (FcγR); genetic polymorphisms of FcγR modify the binding affinity with the Fc of IgG1 (Immunoglobulins Gamma subclass 1). Interestingly, the high-affinity FcγRIIIa (FcγR type IIIa) V/V is associated with increased ADCC in vitro and in vivo. Thus, ADCC could partially account for cetuximab activity. CIFRA is a single arm, open-label, phase II study assessing the activity of cetuximab in combination with irinotecan and fluorouracile in FcγRIIIa V/V patients with KRAS (Kirsten RAt Sarcoma), NRAS (Neuroblastoma Rat Sarcoma), BRAF (B-Rapidly Accelerated Fibrosarcoma) wild type mCRC. The study is designed with a two-stage Simon model based on a hypothetical higher response rate (+10%) of FcγRIIIa V/V patients as compared to previous trials (about 60%) assuming ADCC as one of the mechanisms of cetuximab action. The test power is 95%, the alpha value of the I-type error is 5%. With these assumptions the sample for passing the first stage is 14 patients with >6 responses and the final sample is 34 patients with >18 responses to draw positive conclusions. Secondary objectives include toxicity, responses' duration, progression-free and overall survival. Furthermore, an associated translational study will assess the patients' cetuximab-mediated ADCC and characterize the tumor microenvironment.

The CIFRA study will determine whether ADCC contributes to cetuximab activity in mCRC patients selected on an innovative immunological screening. Data from the translational study will support results'interpretation as well as provide new insights in host-tumor interactions and cetuximab activity.

ELIGIBILITY:
Inclusion Criteria:

* Cytological or histological diagnosis of colorectal adenocarcinoma;
* KRAS, NRAS, BRAF wild-type;
* FcγRIIIaV/V genotype;
* stage IV;
* age <75 years;
* at least 1 measurable lesion;
* ECOG (Eastern Cooperative Oncology Group) Performance Status 0 or 1;
* life expectancy> 3 months;
* negative pregnancy test for all potentially childbearing women;
* written informed consent.

Exclusion Criteria:

* previous systemic anti-tumor treatment (allowed treatment with capecitabine or fluorouracil and radiotherapy in the neoadjuvant setting of rectal tumors with therapy terminated at least 6 months before);
* presence of primary non-treated stenosing colorectal neoplasm;
* neutrophils <2000/mm³ or platelets <100.000/mm³ or hemoglobin <9 g/dl;
* serum creatinine level> 1.5 times the maximum normal value;
* GOT (glutamic oxaloacetic transaminase) and/or GPT (glutamic pyruvic transaminase) >5 times the maximum normal value and/or bilirubin level >3 times the maximum normal value;
* previous malignant neoplasms (excluding basal or spinocellular cutaneous carcinoma or in situ carcinoma of the uterine cervix);
* active or uncontrolled infections;
* other concomitant uncontrolled diseases or conditions contraindicating the study - drugs at clinician evaluation;
* presence of brain metastases;
* refusal or inability to provide informed consent;
* impossibility to guarantee follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-09-05 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Activity | 1 year
  Activity assessed by RECIST criteria version 1.1

SECONDARY OUTCOMES:
Response duration | 1 year
  Time elapsed from date of response to progression occurrence.
Progression-free survival (PFS) | Through study completion, an average of 1 year
  PFS will be determined from the date of treatment start until progression.
Overall survival (OS) | Through study completion, an average of 2 years
  OS will be measured from treatment start until death from any cause.
Toxic effects | At the end of Cycle 1 (each cycle is 14 days)
  Toxic effects assessed by CTCAE of the National Cancer Institute, version 4.0, June 14, 2010

OTHER OUTCOMES:
Percentage of antibody-dependent cell-mediated cytotoxicity (ADCC) in vitro through the evaluation of tumor cell lysis after co-incubation of tumor cells, cetuximab and patient-derived lymphocytes. | Before treatment start
  To study cetuximab-mediated ADCC, peripheral blood mononuclear cells from patients will be isolated, and added in the presence of cetuximab to colorectal cancer cells. The specific cytolysis will be evaluated by sulforhodamine B (SRB) assay and the percentage of lysis will be calculated using the following formula: Cytotoxicity (%) = [1 - (mean test optical density/mean optical density target)] × 100.
Type of cells infiltrating the tumor microenvironment. | Before treatment start
  The primary tissues, and metastases when available, will be characterized for the presence of tumor-infiltrating M1 and M2 macrophages and tumor-infiltrating lymphocytes by immunohistochemistry through the expression of CD163 (ab182422, Abcam), TGF-β (Tumor Growth Factor beta) (ab92486, Abcam), Arginase-1 (GTX113131, Genetex), Osteopontin (ab218237, Abcam], and PD-L1 (Programmed Death-Ligand 1) (E1L3N®, XP®). M1 infiltrating macrophages will be detected through the following antibodies: CD86 (Cluster of Differentiation 86) (ab53004, Abcam), iNOS (inducible Nitric Oxide Synthase) (ab115819, Abcam), IFN-γ (InterFeroN-gamma) (ab218426, Abcam), TNF (Tumor Necrosis Factor) (ab1793, Abcam). Natural Killer (NK) and Cytotoxic T Lymphocytes (CTL) will be characterized as follows: NKP46+ (Clone 195314, R&D system), granzyme B (ab134933, Abcam), Foxp3+ (ab20034, Abcam). Results will be expressed for any type of cells in percentages (numerical proportions of stained cells).

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Nazionale dei Tumori,, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No